CLINICAL TRIAL: NCT05539365
Title: A Phase II Study of Intratumorally Injected Autologous Dendritic Cells (DCs) in PD-L1-Negative Treatment Naïve and in Refractory Metastatic Triple Negative Breast Cancer Patients
Brief Title: Dendritic Cell-Based Treatment Plus Immunotherapy for the Treatment of Metastatic or Unresectable Triple Negative Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never activated.
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 1680021; NCI-2022-07097 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 1680021 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma; Unresectable Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy; Leukapheresis; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ST-alpha-DC1, pembrolizumab) (Experimental): Patients undergo leukapheresis over 90 minutes. Patients then receive ST-alpha-DC1 IT on days 1, 8, and 50 in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab IV on days 8, 29, 50, and 71 in the absence of disease progression or unacceptable toxicity. Patients who are receiving clinical benefit from treatment at the end of day 85, may continue to receive pembrolizumab IV every 3 weeks beyond the 4 study doses. Patients also undergo tumor biopsies on days 1, 8, and 50 and CT scans at baseline and days 50 and 85.
  Interventions: Biological: Alpha-type-1 Polarized Dendritic Cells; Procedure: Biopsy; Procedure: Computed Tomography; Procedure: Leukapheresis; Biological: Pembrolizumab; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Alpha-type-1 Polarized Dendritic Cells — Given IT
  Other Names: alphaDC1
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial tests the safety, side effects, and whether dendritic cell-based treatment and pembrolizumab work in treating patients with triple negative breast cancer that has spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). The term triple-negative breast cancer refers to the fact that the cancer cells don't have estrogen or progesterone receptors (ER or PR) and also don't make any or too much of the protein called HER2 (the cells test "negative" on all 3 tests). Dendritic cell-based treatment works by boosting the immune system (a system in our bodies that protects us against infection) to recognize and destroy the cancer cells. Pembrolizumab, is an immune checkpoint inhibitor drug, that works by targeting molecules that act as a check and balance system for immune responses. Immune checkpoint inhibitor drugs are designed to either "unleash" or "enhance" the cancer immune responses that already exist by either blocking inhibitory molecules or by activating stimulatory molecules. Giving dendritic cell-based therapy and pembrolizumab may decrease symptoms and improve quality of life in patients with triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the clinical efficacy and safety and tolerability of a combination of intratumorally injected autologous dendritic cells (DCs) and pembrolizumab in PD-L1 negative treatment-naive and refractory metastatic triple negative breast cancer patients.

SECONDARY OBJECTIVES:

I. To assess progression-free survival and overall survival in metastatic triple negative breast cancer patients that received the combination of intratumorally injected autologous DCs and pembrolizumab.

II. To assess the clinical efficacy in the non-injected target lesion (optional biopsies for this lesion).

OUTLINE:

Patients undergo leukapheresis over 90 minutes. Patients then receive ST-alpha-DC1 intratumorally (IT) on days 1, 8, and 50 in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab intravenously (IV) on days 8, 29, 50, and 71 in the absence of disease progression or unacceptable toxicity. Patients who are receiving clinical benefit from treatment at the end of day 85, may continue to receive pembrolizumab IV every 3 weeks beyond the 4 study doses. Patients also undergo tumor biopsies on days 1, 8, and 50 and computed tomography (CT) scans at baseline and days 50 and 85.

After completion of study treatment, patients are followed up at 30 and 90 days after the last dose of study drug, and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* Pathologically confirmed diagnosis of unresectable or metastatic triple negative breast cancer (TNBC) with no curative treatment options
* At least 2 target lesions present per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at least one of which is amenable to biopsy and injection
* PD-L1 negative metastatic TNBC patients who are treatment naive in the first linen metastatic setting are eligible
* Both PD-L1 positive and PD-L1 negative metastatic TNBC patients in the second line setting and beyond are eligible
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of =< 2
* Platelets >= 75,000/uL
* Hemoglobin >= 8 g/dL
* Absolute Neutrophil Count (ANC) >= 1500/uL
* Creatinine =< 1.5 x upper limit of normal (ULN) OR creatinine clearance >= 30 mL/min for participant with creatinine levels >1.5 x institutional ULN
* Total bilirubin: =< 2 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 2 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT] =< 3 x institutional ULN (=< 5 x ULN for participants with liver metastases)
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Participants currently treated with systemic immunosuppressive agents, including steroids (> than equivalent of 10 mg daily of prednisone) are ineligible until 3 weeks after removal from immunosuppressive treatment
* Patients with active autoimmune disease or history of transplantation
* Cardiac risk factors including:

  * Patients experiencing cardiac event(s) (acute coronary syndrome, myocardial infarction, or ischemia) within 3 months of signing consent
  * Patients with a New York Heart Association classification of III or IV
* Pregnant or nursing female participants
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=<2 weeks of radiotherapy) to non-CNS disease
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has severe hypersensitivity (>= Grade 3) to pembrolizumab and/or any of its excipients
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has active Human Immunodeficiency Virus (HIV) infection

  * Note: HIV testing is required
* Has active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection

  * Note: Testing for Hepatitis B and Hepatitis C is required
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit comp
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective responses rate (ORR) | Up to 2 years
  Will be assessed by immune related response criteria (iRECIST).
Incidence of adverse events | Up to 30 days after last dose
  Will be assessed using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, and will be summarized by attribution and grade using frequencies and relative frequencies.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  Will be summarized using standard Kaplan-Meier methods, where the median times will be estimated with 90% confidence intervals.
Overall survival (OS) | Up to 2 years
  Will be summarized using standard Kaplan-Meier methods, where the median times will be estimated with 90% confidence intervals.
Objective response rate | Up to 2 years
  Objective response in the target lesion that is not injected will be summarized using frequencies and relative frequencies.

OTHER OUTCOMES:
Health-related quality of life (HR-QOL) | Up to day 85
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) will be summarized by time point (pre- and post-treatment) using the appropriate descriptive statistics. The pre- and post-treatment levels will be compared using a permutation paired t-test.
Quality of Life as measured by the Perceived Stress Scale | Up to day 85
  Measured using validated 10 question "Perceived Stress Scale" which assesses global stress (regardless of source). This 10 question survey uses a 0-4 scale with higher composite score corresponding to greater stress

CONTACTS AND LOCATIONS:
Overall Officials: Shipra Gandhi, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States